CLINICAL TRIAL: NCT02277834
Title: Characterizing the Pancreatic Adenocarcinoma Proteome From Pancreatic Juice
Brief Title: Characterizing the Pancreatic Cancer Proteome From Pancreatic Juice
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: UAB 1361
Record Dates: First submitted 2014-10-06; First posted 2014-10-29 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples will be in 3 differant cohorts;
  1. Subject with biopsy-proven Pancreatic Adenocarcinoma of the pancreas
  2. Subjects witha diagnosis of Pancreatitis
  3. Subject with NO pancreatic abnormality
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- pancreatic adenocarcinoma: 15 patients receiving Endoscopic Retrograde Cholangiopancreatography with suspected pancreatic adenocarcinoma (localized or metastatic).
- chronic pancreatitis: 15 patients with a history of chronic pancreatitis that are having Endoscopic Retrograde Cholangiopancreatography .
- non-pancreatic, non-neoplastic disorders: 15 patients undergoing an Endoscopic Retrograde Cholangiopancreatography for non-pancreatic, non-neoplastic indications.

SUMMARY:
Currently, X-rays and blood tests often miss pancreatic cancer. In this study, we are collecting and studying the fluid produced by the pancreas as a way to detect pancreatic cancer at an earlier stage.

DETAILED DESCRIPTION:
Pancreatic cancer is very difficult to detect and treat, and patients with this cancer generally live fewer years than patients with other types of cancer. Part of the reason why pancreatic cancer is so hard to treat is because it is usually discovered when it is too advanced to be able to treat. The goal of this protocol is to find a way to detect pancreatic cancer earlier, when it is still treatable in order to improve the survival of patients.

The pancreas is a gland which produces digestive juices that mix with food in the intestines. Normal patients as well as patients with pancreatic cancer produce these juices. Other researchers have collected this fluid from very small numbers of patients and their results suggest that pancreatic fluid can be used to detect pancreatic cancer. One of the major issues with these results is that pancreatic fluid from only a very few number of patients has been collected and analyzed. In order to find out whether the pancreatic fluid can be used as a standard test for pancreatic cancer, the fluid from a greater number of patients needs to be analyzed. Also, of all the different chemicals in the pancreatic fluid, in this study we will try to figure out what the most important chemicals are in diagnosing pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:Group A:

1. Male or females that have suspected pancreatic adenocarcinoma, localized or metastatic.
2. The pancreatic adenocarcinoma must be active, with active intra-pancreatic tumor documented within the last 3 months by CT or MRI scan.
3. At least 19 years of age. (All Cohorts)
4. In the Investigator's judgment, participant is mentally competent to provide informed consent to participate in the study. (All Cohorts)
5. Eastern Cooperative Oncology Group(ECOG) performance status of 0-2. (All Cohorts)
6. Negative urine pregnancy test at screening, if applicable. (All Cohorts)
7. The patient must already have a completed, active consent for either endoscopic ultrasound(EUS) and/or endoscopic retrograde cholangiopancreatography (ERCP) at University of Alabama at Birmingham(UAB). (All Cohorts)

Group B:

1. Male or female patients that have had chronic pancreatitis for at least 6 months.
2. CT abdomen or MRI abdomen within the last 3 months demonstrating no suspicion of pancreatic adenocarcinoma.

Group C:

1.Male or female patients already scheduled to undergo upper endoscopy for non-pancreatic, non-neoplastic indications.

Exclusion Criteria:Group A:

1. The participant is medically unfit to undergo upper endoscopy.
2. No cancer-directed therapy administered within the last 3 months. This includes any of the following: surgical resection, chemotherapy, radiation therapy, immunologic or biologic therapy.
3. Participants with a known allergy to secretin.
4. Participants who are pregnant or lactating, or intending to become pregnant during the study.
5. Participants of childbearing potential who refuse a pregnancy test.
6. Participants who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
7. Participants who have participated in an investigational surgical, drug, or device study within the past 30 days.
8. Participants who currently have a biliary stent in place.
9. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
10. The endoscopic pancreatic biopsy does not show adenocarcinoma.

Group B:

1. The participant is medically unfit to undergo upper endoscopy.
2. The participant has a suspicion of pancreatic adenocarcinoma on imaging within the last 3 months.
3. Participants with a known allergy to secretin.
4. Participants who are pregnant or lactating, or intending to become pregnant during the study.
5. Participants of childbearing potential who refuse a pregnancy test.
6. Participants who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
7. Participants who have participated in an investigational surgical, drug, or device study within the past 30 days.
8. Participants who currently have a biliary stent in place.
9. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.

Group C:

1. The participant is medically unfit to undergo upper endoscopy.
2. The participant has a history of, or current clinical suspicion of pancreatic adenocarcinoma or pancreatitis.
3. The participant has a history of any type of gastrointestinal malignancy within the last 5 years.
4. Participants with a known allergy to secretin.
5. Participants who are pregnant or lactating, or intending to become pregnant during the study.
6. Participants of childbearing potential who refuse a pregnancy test.
7. Participants who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
8. Participants who have participated in an investigational surgical, drug, or device study within the past 30 days.
9. Participants who currently have a biliary stent in place.
10. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.

    -

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group A: Participants with a confirmed diagnosis of a pancreatic adenocarcinoma will be enrolled in this study. Potential participants will be identified from the Surgical Oncology and Gastroenterology outpatient settings.
  Group B: Participants with a confirmed diagnosis of chronic pancreatitis will be enrolled in this study. Participants will be derived from the Gastroenterology and Gastrointestinal Surgery outpatient setting.
  Group C: Participants undergoing endoscopy for non-pancreatic, non-neoplastic indications. The typical patient population we anticipate recruiting to this group with be those with non-malignant, non-pancreatitis biliary calculous disease. Participants will be derived from the Gastroenterology outpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Compare the proteomic signature of pancreatic adenocarcinoma , pancreatic cancer and control participants to the disease process | 120 months from First subject enrolled
  Characterization of the proteomic signature of patients with pancreatic adenocarcinoma, pancreatic cancer, and control participants. This will be accomplished by classifying a group or set of similar proteomic profiles(once we(once we have developed from the samples obtained a list of known proteomic profiles taht are found in all pancreatic adenocarcinoma subjects) that are specific to the disease process,of pancreatic adenocarcinoma.

SECONDARY OUTCOMES:
Compare the proteomic profile between pancreatic cancer and pancreatitis | 120 months from First subject enrolled
  Using the discovered pancreatic adenocarcinoma proteomic profile we will differentiate a documentable difference from pancreatic cancer and pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Carlo M Contreras, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No